CLINICAL TRIAL: NCT05932914
Title: Liver Biopsy Following Gene Therapy For Hemophilia
Status: Not yet recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Methodist University Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: LIVBX
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: AAV-mediated factor VIII (FVIII) gene transfer; AAV-mediated factor IX (FIX) gene transfer; Gene Therapy; Hemophilia A; Hemophilia B; Transjugular liver biopsy
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Those who meet the Eligibility Criteria
  Interventions: Procedure: Liver Biopsy

INTERVENTIONS:
Procedure: Liver Biopsy — Standard transjugular liver biopsy under moderate sedation

SUMMARY:
This observational study will obtain liver biopsy samples and evaluate the long-term effect of adeno-associated virus (AAV)-mediated gene therapy on the liver tissue in adult patients with hemophilia A or hemophilia B who have previously been treated with a factor VIII or factor IX gene-containing AAV-vector for liver-targeted gene transfer. Participants are from a cohort of patients treated with AAV-mediated gene transfer and at least 6 months after vector infusion.

DETAILED DESCRIPTION:
This is a prospective cohort study evaluating the effect of AAV-mediated gene therapy on the liver in adult patients with hemophilia A or hemophilia B who have previously been treated with a FVIII/FIX gene-containing AAV-vector for liver-targeted gene transfer.

To better understand the effect of AAV-mediated gene transfer on the liver, eligible participants can allow the use and analysis of already existing liver tissue samples, taken and preserved after having received gene therapy. Alternatively, eligible participants can consent to providing a new liver tissue sample which will be obtained by undergoing a standard transjugular liver biopsy (TJLB) procedure under moderate sedation. . The procedure will be done as outpatient (day 1) with post procedure follow-up on day 2, 3, 4 and 14.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to 80 years
* Patients, who were enrolled and treated in one of the following clinical trials:

  * AGT4HB (EudraCT number: 2005-005711-17; NCT00979238) - FIX AAV gene therapy trial (sponsor: St. Jude Children's Research Hospital)
  * GO8 (EudraCT number:2014-003880-38; NCT02576795) - FVIII AAV gene therapy trial (sponsor: University College, London)
* Able to give informed consent
* Able to comply with study requirements

Exclusion Criteria (Do not apply to participants who will not undergo liver biopsy, and have leftover liver tissue from a previous biopsy procedure, because all exclusion criteria only cover the safety considerations for the biopsy procedure.):

* Any condition that, in the opinion of the investigator or sponsor of the ongoing clinical trial in which the patient is participating in, would prevent the patient from fully complying with the requirements of the clinical trial and/or would influence or interfere with evaluation and interpretation of subject safety or efficacy result of that ongoing clinical trial
* Platelet count <140x10^9/L
* INR >1.5
* Abnormal kidney function with estimated GFR <50 mL/min (calculated using the CKD-EPI equation)
* Known allergy to iodine-based intravenous contrast agents
* Known allergy to local or general anesthetics
* Known allergic reaction to FVIII/FIX concentrate infusions
* Presence of FVIII inhibitor or FIX inhibitor (historical result can be used if done within 14 weeks of this liver biopsy)
* Evidence of any bleeding disorder other than hemophilia A or B

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who meet the Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the number of hepatocytes transduced with AAV vector genome in liver biopsy samples analyzed by FISH | single time point (day of biopsy)
  Fluorescence in situ hybridization (FISH)

SECONDARY OUTCOMES:
The degree of hepatocyte damage at a morphological level | single time point (day of biopsy)
  Standard and immunohistochemical tissue staining
The number and type of hot spots for integration of AAV provirus in liver cells | single time point (day of biopsy)
  DNA sequencing
The number of hepatocytes revealing FVIII/FIX RNA in-situ transcripts | single time point (day of biopsy)
  Assessment of RNA in-situ transcripts
The number and types of epigenetic changes within the AAV genome in the liver | single time point (day of biopsy)
  DNA methylation analysis and histone association studies
The qualitative and quantitative assessment of the RNA transcriptome | single time point (day of biopsy)
  Assessment of RNA transcriptome

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Reiss, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols